CLINICAL TRIAL: NCT03911011
Title: Gas Diffusion in and Out of an Air Pocket After a Simulated Snow Avalanche and Its Impacts on Human Physiological Parameters.
Brief Title: Physiological Values When Breathing in an Air-pocket. Mountain Lab 2019 (ML2019)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Ullevaal University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018/2478
Record Dates: First submitted 2019-02-22; First posted 2019-04-10 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Accident Caused by Snow Avalanche
Keywords: avalanche, survival, physiology

STUDY DESIGN:
Intervention Model Description: A field study designed as a crossover clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fresh air (Active Comparator): 2 litres of fresh air
  Interventions: Other: Fresh air
- no fresh air (No Intervention): no supply of fresh air

INTERVENTIONS:
Other: Fresh air — Fresh air insufflation of 2 L/min toward mouth/nose.
  Arms: Fresh air

SUMMARY:
The literature describes and report neurologic intact patients surviving an avalanche several hours after they were buried. The most important factor for surviving more than 15-35 min of burial is considered to be the presence of an air-filled space around the head and neck, termed an air pocket. Little is known how the inspired air is influenced by the patients breathing and how oxygen and carbon dioxide diffuse through snow.

DETAILED DESCRIPTION:
In a controlled and simulated avalanche scenario the investigators want to investigate how oxygen (O2) and carbon dioxide (CO2) diffuse and how rebreathing of CO2 in addition to mild hypoxia influence standardized physiological parameters in two scenarios: Fresh air and no fresh air delivered into the air pocket. The project is a field study designed to measure and document gas diffusion through snow. The outcome measures are: (1) Concentration of O2 and CO2 in the air pocket and 50 cm from the pocket. (2) Time interval for development of threshold values for concentration of O2 and CO2. The investigators will also monitor physiologic measures such as: Electrocardiogram (ECG), continuous invasive blood pressure, cerebral oximetry, continuous pulse oximetry, transthoracic impedance, and gas content in expired air. Subjective evaluation of comfort will also be scored. Twenty healthy young volunteers with written consent to participate will be used as test subjects.

The study may have a clinical consequence for better outcome, for victims of avalanches by providing additional air or oxygen close to the patient. The study will also measure specific body measures and spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be Healthy
* Subject must be non smoking
* Subject must have normal BMI

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Time | 25 minutes
  Time to reaching a threshold of physiology parameters or time limit

OTHER OUTCOMES:
Physiology | 25 minutes
  Values of Physiology parameters

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Klausen, PhD, Study Director — Director, Department for Anaesthesia and Intensive Care
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No